CLINICAL TRIAL: NCT04661735
Title: Retrospective Analysis - Scoring Systems in Intensive Care Medicine
Brief Title: Intensive Care Unit Risk Score
Acronym: ICURS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Felix Balzer, MD, MSc., PhD, Professor, Charite University, Berlin, Germany
Other Study IDs: ICURS
Record Dates: First submitted 2020-12-04; First posted 2020-12-10 (Actual); Last update posted 2023-09-08 (Actual); Status verified 2023-09

CONDITIONS: Mortality in Intensive Care Units; Complications Infection; Alarm Fatigue
Keywords: scores; intensive care unit; patient monitoring; alarm management
MeSH Terms: conditions — Alert Fatigue, Health Personnel

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Subject of the planned project is the retrospective analysis of routine data of digital patient files of the Department for Anaesthesiology and Surgical Intensive Care Medicine, to test whether the predictive values of intensive care scoring systems with regard to perioperative mortality and morbidity can be improved by continuous score calculation and by using machine learning and time series analysis methods.

DETAILED DESCRIPTION:
A scoring system usually consists of two parts - a score (a number reflecting the severity of the disease) and a probability model (equation indicating the probability of an event, e.g. the death of the patient in hospital). Scoring systems have been used in intensive care medicine for decades and can help to assess the effectiveness of treatment or identify comparable patients for study purposes. Scoring systems that are used in intensive care medicine are for example

* Acute Physiology, Age, Chronic Health Evaluation II (APACHE II)
* Simplified Acute Physiology Score II (SAPS II)
* Multiple Organ Dysfunction Score (MODS)
* Sequential Organ Failure Assessment (SOFA)
* Logistic Organ Dysfunction System (LODS)
* MPM II-Admission (Mortality Probability Models (MPM II)
* Organ Dysfunction and Infection score (ODIN)
* Three-Day Recalibrating ICU Outcomes (TRIOS)
* Glasgow coma score (GCS)
* Discharge Readiness Score (DRS) The above-mentioned scoring systems are already being collected regularly in the respective hospital's departments. In a recent study by Badawi et al. it could be shown that scoring systems allow more accurate predictions when calculated continuously. However, due to the patient collectives investigated, these results can only be transferred to other patient groups to a limited extent. Furthermore, only the scoring systems APACHE, SOFA and DRS were analyzed.

Therefore, in the present study, all of the above scoring systems will be calculated continuously (once per minute) using routine data from the digital patient records and optimized by applying machine learning and methods of time series analysis.

On the anesthesiologically managed intensive care units of the respective hospital, there is no campus-wide standard with regard to alarm management. Accordingly, we estimate the rate of alarm fatigue (ignoring alarms due to many false alarms) to be very high. In order to optimize the alarm management, alarms from the patient monitoring devices will be evaluated retrospectively and combined with the data mentioned above to determine, for example, whether more frequent alarms are to be expected for certain types of diseases (e.g. sepsis), or scores (e.g., high APACHE score) and how the alarm limit setting can be optimized.

ELIGIBILITY:
Inclusion Criteria:

- Patients with admission between 01.01.2006 and 30.09.2023

Exclusion Criteria:

* Patients under 18 years of age.
* Incomplete patient records.
* Intensive stay of less than 24 hours.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Age from 18 years. The respective intensive care department carries out approximately 5000 intensive care treatments per year on persons of each sex.
Sampling Method: Non-Probability Sample
Enrollment: 60000 (Estimated)
Dates: Start 2006-01-01 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Prediction of patient outcome | 2006 - 2023
  Identification of scores with a high on impact mortality, complications and length of stay in the intensive care unit

SECONDARY OUTCOMES:
Predictive model for alarm load | 2020 - 2023
  Identification of items leading to a high alarm load measured by number of alarm per day per bed in the intensive care unit
Predictive model for actionable alarms | 2020 - 2023
  Identification of items leading to a high number of actionable alarms measured by number of actionable alarms per day per bed in the intensive care unit

CONTACTS AND LOCATIONS:
Overall Officials: Felix Balzer, Prof, Principal Investigator — Charite University, Berlin, Germany
Locations (1):
- Charite Universtitaetsmedizin, Berlin, Germany